CLINICAL TRIAL: NCT03971799
Title: Phase 1/2 Study of Anti-CD33 Chimeric Antigen Receptor-Expressing T Cells (CD33CART) in Children and Young Adults With Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Study of Anti-CD33 Chimeric Antigen Receptor-Expressing T Cells (CD33CART) in Children and Young Adults With Relapsed/Refractory Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Center for International Blood and Marrow Transplant Research (Network)
Collaborators: National Marrow Donor Program (Other); St. Baldrick's Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-CD33CART
Record Dates: First submitted 2019-05-29; First posted 2019-06-03 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Acute Myelogenous Leukemia
Keywords: CD33CART cells; Children/young adults
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: A 3+3 dose escalation design will be used to determine maximum tolerated dose for both autologous and allogeneic recipients in Phase 1 and Simon's two-stage design will be used to evaluate the efficacy of CD33CART in Phase 2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- CD33CART autologous (Experimental): Patients who receive an autologous CD33CART cell infusion
  Interventions: Biological: CD33CART autologous
- CD33 CART allogeneic (Experimental): Patients who receive an allogeneic CD33CART cell infusion
  Interventions: Biological: CD33CART allogeneic

INTERVENTIONS:
Biological: CD33CART autologous — The treatment regimen will consist of lymphodepleting (LD) chemotherapy followed by autologous CD33CART infusion:
  LD option #1 (IV fludarabine 25 mg/m2/dose administered Days -4 to -2 and IV cyclophosphamide 900 mg/m2/dose on Day -2) or LD option #2 (IV fludarabine 30 mg/m2 on days -5, -4, -3, and -2; and IV cyclophosphamide 500 mg/m2 on days -3 and -2).
  Subjects will then proceed to allogeneic HCT or alternative therapy as clinically applicable.
  Arms: CD33CART autologous
Biological: CD33CART allogeneic — The treatment regimen will consist of lymphodepleting (LD) chemotherapy followed by allogeneic CD33CART infusion:
  LD option #1 (IV fludarabine 25 mg/m2/dose administered Days -4 to -2 and IV cyclophosphamide 900 mg/m2/dose on Day -2) or LD option #2 (IV fludarabine 30 mg/m2 on days -5, -4, -3, and -2; and IV cyclophosphamide 500 mg/m2 on days -3 and -2).
  Subjects will then proceed to allogeneic HCT or alternative therapy as clinically applicable.
  Arms: CD33 CART allogeneic

SUMMARY:
This phase 1/2 trial aims to determine the safety and feasibility of antiCD33 chimeric antigen receptor (CAR) expressing T cells (CD33CART) in children and adolescents/young adults (AYAs) with relapsed/refractory acute myeloid leukemia (AML). The trial will be done in two phases: Phase 1 will determine the maximum tolerated dose of CD33CART cells using a 3+3 trial design, with dose-escalation for autologous products separated from dose-escalation for an allogeneic arm. Phase 2 is an expansion phase designed to evaluate the rate of response to CD33CART.

DETAILED DESCRIPTION:
This study consists of two phases. The objectives of Phase 1 and Phase 2 are:

Phase 1:

Autologous Arm: To determine the maximum tolerated dose of lentivirally transduced autologous CD33-redirected CAR-T cells (CD33CART) in children and young adults with relapsed/refractory AML

Allogeneic Arm: To determine the maximum tolerated dose of lentivirally transduced allogeneic CD33-redirected CAR-T cells (ALLO-CD33CART) in children and young adults with post-HSCT relapsed/refractory AML

Phase 2:

To determine the percentage of recipients treated with CD33CART who achieve morphologic remission (<5% blasts in marrow) at Day 28 post-CD33CART cell infusion

ELIGIBILITY:
Recipients >1 year to <35 years of age with AML in 2nd or greater relapse or refractory to 2 or more induction attempts without central nervous system (CNS) CNS3 disease and who have a suitable allogeneic HCT donor and a performance status of > 50% may be eligible for study. For those patients with post-HCT relapse enrolled to the allogeneic arm, patients must be at least 100 days post-HCT and not have any evidence of active GVHD or be on systemic immunosuppression for the GVHD.

Related Donors: A donor from prior HCT who is fully matched by institutional standards and able to undergo apheresis for T-cell collection.

Recipient Inclusion Criteria

1. Recipients must have CD33+ AML in second or greater relapse, post-transplant relapse, or have demonstrated chemotherapy-refractory disease (definitions in criteria 2c) to be eligible to participate in this trial.
2. Disease status at the time of enrollment:

   1. Recipients in second or greater relapse will be eligible with relapse defined as >5% blasts (bone marrow) after second documented complete remission
   2. Any degree of detectable disease post-transplant relapse will be eligible (with flow cytometric confirmation of CD33+ myeloid leukemia of at least 0.1%)
   3. Refractory disease is defined as persistent bone marrow involvement with >5% blasts after two courses of induction chemotherapy for patients at initial presentation or >5% bone marrow blasts after one course of re-induction chemotherapy for patients in relapse;
3. CD33 expression must be detected on greater than 50% of the malignant cells by immunohistochemistry or greater than 80% by flow cytometry;
4. Age: Greater than or equal to 1 year of age and less than or equal to 35 years of age at time of enrollment.
5. All recipients must have an allogeneic HCT donor identified with a plan to proceed to HCT conditioning within 6-8 weeks of CD33CART cell infusion;
6. Patients with two prior allogenic donor stem cell transplants must be medically fit for a third allogenic donor stem cell transplant
7. Performance status: > 50% (for recipients > 16 years of age use Karnofsky ≥ 50%; recipients < 16 years of age: Lansky scale ≥ 50%) (see Appendix II). Recipients who are unable to walk because of paralysis, but who are upright in a wheelchair will be considered ambulatory for the purpose of calculating the performance score;
8. Adequate organ function as defined by:

   1. Cardiac function: left ventricular ejection fraction (LVEF) ≥ 45% or fractional shortening ≥28%
   2. Pulmonary function: baseline oxygen saturation > 92% on room air at rest
   3. Hepatic function:

      * Total bilirubin < grade 2 bilirubin CTCAE version 5 (<3 x ULN) (except in case of recipients with documented Gilbert's disease > 3 x ULN)
      * AST (SGOT)/ALT (SGPT) < 5 x institutional ULN (< grade 3)
   4. Renal function: Serum creatinine must be < 1.2 x institutional upper limit of normal (ULN) according to age. If the serum creatinine is greater than 1.2 x ULN, the patient must have a creatinine clearance (CrCl) > 70mL/min/1.73 m2 (measured by 24 hour- urine specimen or radioisotope GFR).
9. Recipients > 18 years of age must have the ability to give informed consent according to applicable regulatory and local institutional requirements. Legal guardian permission must be obtained for recipients < 18 years of age. Pediatric recipients will be included in age-appropriate discussion in order to obtain assent; Adults with cognitive impairment who are unable to consent and those with Down Syndrome are also eligible for this protocol with the proper assessments as outlined in Protocol Section 11.2.
10. Enrollment in the NMDP protocol: Protocol for a Research Database for Hematopoietic Cell Transplantation, Other Cellular Therapies and Marrow Toxicity Injuries.

Recipient Exclusion Criteria

Recipients meeting any of the following criteria are not eligible for participation in the study:

1. Recipients with radiologically-detected CNS chloromas or CNS 3 disease (presence of ≥ 5/μL white blood cells (WBCs) in cerebral spinal fluid (CSF) and cytospin positive for blasts [in the absence of a traumatic lumbar puncture] and/or clinical signs of CNS leukemia such as a cranial nerve palsy from active disease). Recipients with adequately treated CNS leukemia are eligible;
2. Hyperleukocytosis (≥ 50,000 blasts/μL) or rapidly progressive disease that in the estimation of the investigator and sponsor would compromise ability to complete study therapy;
3. Pregnancy (negative serum or urine pregnancy test must be obtained at time of enrollment for females of childbearing potential and to be repeated 72 hours prior to lymphodepleting chemotherapy regimen);
4. Breast feeding;
5. Sexually active female recipients of childbearing potential and male recipients who are of childbearing potential and are unwilling to practice birth control at time of enrollment and for four months after receiving the lymphodepletion preparative regimen;
6. Active or uncontrolled viral, bacterial or fungal infection. May be receiving ongoing therapy for controlled infection
7. Recent prior therapy:

   1. At treatment enrollment:

      Patients may be on lower-intensity chemotherapy (e.g., TKIs, venetoclax, hydroxyurea, azacytidine, decitabine or similar agents) at the time of enrollment to prevent disease progression. There is no timing restriction of intrathecal chemotherapy for enrollment.
   2. Prior to apheresis: The following wash-out periods apply prior to apheresis

      * Systemic chemotherapy ≤ 14 days with the exception of:

        * Hydroxyurea: 1 day
        * Azacytidine/decitabine and/or venetoclax: 7 days
      * Intrathecal chemotherapy > 3 days
      * Tyrosine kinase inhibitors: 3 half-lives or 7 days, whichever is shorter (See Appendix XVIII)
      * Checkpoint inhibitors or antibody-based therapies: 3 half-lives
      * Investigational anti-neoplastic agents: 28 days
      * Clofarabine or nitrosureas: 42 days
      * Steroid therapy: Not allowed unless at or below physiologic doses (eg, hydrocortisone replacement for prior adrenal insufficiency)
      * Radiation therapy: Radiation therapy (including CNS) must have been completed at least 21 days prior to apheresis with the exception of no time restriction if the volume of bone marrow treated is less than 10% and also the recipient has measurable/evaluable disease outside the radiation field.
      * CAR T-cell therapy: Excluded unless at least 30 days from prior CAR T-cell infusion and without detectable circulating CAR T-cells **Please see protocol section 2.5.1 for guidance on wash-out parameters prior to initiation of LD chemotherapy
8. Recipients with any history of allogeneic stem cell transplantation are excluded if:

   1. Recipients are less than 100 days post-transplant OR
   2. Recipients have evidence of ongoing active GVHD and are taking immunosuppressive agents (>0.5 mg/kg/methylprednisolone equivalents or other immunosuppression for GVHD treatment) OR
   3. Recipients have received DLI within 30 days prior to enrollment OR
   4. Recipients are on active immunosuppression for GVHD prophylaxis (must be off for 30 days prior to enrollment)
   5. Recipients who enroll to the ALLO-CD33CART arm must not have had any prior history of > grade 3 acute GVHD or severe chronic GVHD
9. HIV/HBV/HCV Infection:

   1. Seropositive for HIV 1 or 2 (Recipients with HIV are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in recipient receiving combination antiretroviral therapy in the future should study results indicate effectiveness)
   2. Seropositive for Hepatitis C or positive for Hepatitis B surface antigen (HbsAG)
10. Uncontrolled, symptomatic, intercurrent illness including but not limited to infection, congestive heart failure, unstable angina pectoris, cardiac arrhythmia, psychiatric illness, or social situations that would limit compliance with study requirements or in the opinion of the site PI would pose an unacceptable risk to the recipient
11. Active second malignancy will not be eligible with the following exceptions:

    1. Treatment-related or secondary CD33+ myeloid malignancy which may potentially benefit from CD33CART (which may be considered for enrollment),
    2. Carcinoma in situ of the cervix (which may be considered for enrollment),
    3. Recipient is in remission from a prior second malignancy (which may be considered for enrollment)
12. History of severe, immediate hypersensitivity reaction attributed to compounds of similar chemical or biologic composition to any agents used in study or in the manufacturing of the cells (i.e. gentamicin).

Donor inclusion criteria

1. Must be the same donor whose cells were used as the source for the patient's most recent stem cell transplant
2. Donors > 18 years of age must have the ability to give informed consent according to applicable regulatory and local institutional requirements. Legal guardian permission must be obtained for donors < 18 years of age. Pediatric donors will be included in age-appropriate discussion in order to obtain assent;
3. HLA-matched related sibling (or alternative fully matched relative)
4. Adequate venous access for peripheral apheresis, or without a contradiction to undergoing temporary line placement.

   1. For donors who have previously undergone collection for DLI and have a cryopreserved unmobilized product, this may be considered for use as the starting material

Donor exclusion criteria

1. Pregnancy (negative serum or urine pregnancy test must be obtained at time of enrollment for females of childbearing potential and to be repeated 72 hours prior to apheresis)
2. HIV/HBV/HCV Infection:

   1. Seropositive for HIV 1 or 2
   2. Seropositive for Hepatitis C or positive for Hepatitis B surface antigen (HbsAG)
3. Uncontrolled, symptomatic, intercurrent illness including but not limited to infection, congestive heart failure, unstable angina pectoris, cardiac arrhythmia, psychiatric illness, or social situations that would limit compliance with study requirements or in the opinion of the site PI would pose an unacceptable risk to the donor

Ages: 1 Year to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Estimated)
Dates: Start 2020-01-08 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2039-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose - Autologous Arm | Day 28 post CD33CART infusion
  To determine the maximum tolerated dose of lentivirally-transduced autologous CD33-redirected CAR-T cells (CD33CART) in children and young adults with relapsed/refractory AML
Maximum tolerated dose - Allogeneic Arm | Day 28 post CD33CART infusion
  To determine the maximum tolerated dose of lentivirally-transduced allogeneic CD33-redirected CAR-T cells (ALLO-CD33CART) in children and young adults with post-HSCT relapsed/refractory AML
Morphologic remission | Day 28 post CD33CART infusion
  To determine the percentage of recipients treated with CD33CART who achieve morphologic remission (<5% blasts in marrow) at Day 28 post-CD33CART cell infusion

SECONDARY OUTCOMES:
Feasibility of CD33CART manufacture | 2 weeks post start of CD33CART manufacture
  To determine the feasibility of manufacturing CD33CART for recipients with AML
Feasibility of CD33CART infusion | 6 weeks post apheresis
  To determine the feasibility of infusing CD33CART in recipients with AML
Molecular Cytokine release syndrome (CRS), sinusoidal occlusion syndrome (SOS), or other CD33CART related toxicities | 8 weeks post CD33CART infusion
  To determine the incidence and severity of cytokine release syndrome (CRS), sinusoidal occlusion syndrome (SOS), or other CD33CART related toxicities
Overall survival, event-free survival and treatment-related mortality | 28 days post CD33CART infusion
  To estimate the overall survival, event-free survival, and treatment-related mortality at Day 28 post-CD33CART
Morphologic remission | 28 days post CD33CART infusion
  To determine the percentage of recipients treated with CD33CART who achieve morphologic remission (<5% blasts in marrow) at Day 28 post-CD33CART cell infusion (for those in Phase I)
Molecular remission | 28 days post CD33CART infusion
  To determine the percentage of recipients treated with CD33CART who achieve molecular remission (for those with an identified molecular marker) at Day 28 post-CD33CART cell infusion
MRD negativity | 28 days post CD33CART infusion
  To determine minimal residual disease [MRD] negativity by flow cytometry (<0.1%) at Day 28 post-CD33CART cell infusion
GVHD | 30 days post CD33CART infusion
  To determine the incidence and severity of acute graft-versus-host disease (GVHD) in patients treated on the allogeneic arm (ALLO-CD33CART).
Allogeneic hematopoietic stem cell transplantation | 6 weeks post CD33CART infusion
  To determine the percentage of recipients able to proceed to allogeneic hematopoietic stem cell transplantation following treatment with CD33CART
SOS and other post-transplant toxicities | 6 weeks post HCT
  For treatment population that subsequently proceeds to HSCT: To determine the percentage of recipients able to proceed to allogeneic hematopoietic stem cell transplantation following treatment with CD33CART
Post-HCT time to engraftment | 6 weeks post HCT
  For treatment population that subsequently proceeds to HSCT: To evaluate the post-HCT time to engraftment, transplant related mortality, incidence of acute and chronic graft-versus-host disease (aGVHD and cGVHD).

CONTACTS AND LOCATIONS:
Overall Officials: Nirali Shah, MD, MHSc, Principal Investigator — National Cancer Institute (NCI); Richard Aplenc, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (6):
- United States (6):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - National Cancer Institute - NIH, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Seattle Children's Hospital/Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qin H, Yang L, Chukinas JA, Shah N, Tarun S, Pouzolles M, Chien CD, Niswander LM, Welch AR, Taylor N, Tasian SK, Fry TJ. Systematic preclinical evaluation of CD33-directed chimeric antigen receptor T cell immunotherapy for acute myeloid leukemia defines optimized construct design. J Immunother Cancer. 2021 Sep;9(9):e003149. doi: 10.1136/jitc-2021-003149. PMID 34531250
- See also: Anti-CD22 Chimeric Antigen Receptor (CAR) T Cells in Children and Young Adults With Recurrent or Refractory CD19/CD22-expressing B Cell Malignancies — https://clinicaltrials.gov/ct2/show/NCT02315612?term=CD22+nirali+shah&rank=1
- See also: CD19/CD22 Chimeric Antigen Receptor (CAR) T Cells in Children and Young Adults With Recurrent or Refractory CD19/CD22-expressing B Cell Malignancies — https://clinicaltrials.gov/ct2/show/NCT03448393?term=CD22+nirali+shah&rank=2